CLINICAL TRIAL: NCT03778554
Title: Danish Trial of Beta Blocker Treatment After Myocardial Infarction Without Reduced Ejection Fraction (DANBLOCK)
Brief Title: Danish Trial of Beta Blocker Treatment After Myocardial Infarction Without Reduced Ejection Fraction
Acronym: DANBLOCK
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Amager Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other); Bornholm Hospital (Unknown); Gentofte Hospital (Unknown); Glostrup University Hospital, Copenhagen (Other); Herlev Hospital (Other); Hvidovre University Hospital (Other); Nordsjaellands Hospital (Other); Holbaek Hospital (Unknown); Nykoebing Hospital (Unknown); Naestved Hospital (Other); Zealand University Hospital (Other); Slagelse Hospital (Other); Odense University Hospital (Other); Svendborg Hospital (Other); Sydvestjysk Sygehus (Unknown); Hospital of Southern Jutland (Other); Sygehus Lillebaelt (Vejle and Kolding) (Unknown); Aarhus University Hospital (Other); Hospitalsenheden Midt (Unknown); Hospitalsenheden Vest (Other); Regionshospitalet Horsens (Other); Silkeborg Sygehus (Unknown); Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Eva Prescott, Professor, MD, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-002699-42; 2018-002699-42 (EudraCT Number)
Record Dates: First submitted 2018-12-10; First posted 2018-12-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction; Non-ST Elevation Myocardial Infarction (nSTEMI); ST Elevation Myocardial Infarction
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction | interventions — Metoprolol; Bisoprolol; Carvedilol; Nebivolol

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled, open-label, blinded endpoint (PROBE design)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta blocker treatment (Experimental): Treatment with beta blockers plus standard of care. Type and dosage according to treating cardiologist choice
  * Bisoprolol up to a total dose of 10 mg daily
  * Carvedilol up to a total dose of 50 mg daily
  * Metoprolol succinate up to a total dose of 200 mg daily
  * Nebivolol up to a total dose of 10 mg daily
  Interventions: Drug: Metoprolol Succinate; Drug: Bisoprolol; Drug: Carvedilol; Drug: Nebivolol
- No beta blocker treatment (No Intervention): Standard care without beta blocker treatment

INTERVENTIONS:
Drug: Metoprolol Succinate — Eligible patients randomized to receive long-term therapy with oral beta-blockade
  Arms: Beta blocker treatment
Drug: Bisoprolol — Eligible patients randomized to receive long-term therapy with oral beta-blockade
  Arms: Beta blocker treatment
Drug: Carvedilol — Eligible patients randomized to receive long-term therapy with oral beta-blockade
  Arms: Beta blocker treatment
Drug: Nebivolol — Eligible patients randomized to receive long-term therapy with oral beta-blockade
  Arms: Beta blocker treatment

SUMMARY:
To determine whether long-term treatment with oral betablocker therapy after myocardial infarction in patient with no heart failure reduces the composite outcome of recurrent MI, all-cause mortality, revascularisation with percutaneous coronary intervention or coronary artery bypass graft, ischemic stroke, incident heart failure, or malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin.

DETAILED DESCRIPTION:
Aim: To determine whether long-term treatment with oral betablocker (BB) therapy after myocardial infarction (MI) in patient with no heart failure reduces the composite outcome of recurrent MI, all-cause mortality, revascularisation with percutaneous coronary intervention or coronary artery bypass graft, ischemic stroke, incident heart failure, or malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin.

The inclusion- and event rate in DANBLOCK have been continuously assessed since the first patient was randomized in December 2018. The inclusion- and event rate have been lower than expected, in part due to COVID-19. To enhance feasibility, the decision was made by the Steering Committees to combine the data from DANBLOCK with the data from the Norwegian BETAMI (NCT03646357) and publish the primary endpoint, key secondary endpoints and most other secondary endpoints together (presented below).

The trials have similar designs, only minor differences in study entry criteria, and were, from the very beginning, coordinated with the aim of conducting sub-studies on pooled data. The primary endpoint has been harmonized without knowledge of the distribution of events. BETAMI and DANBLOCK will remain separate trials until the end of follow-up, where data from the trials will be combined and main results published together.

Intervention: BB therapy versus no therapy.

Main Inclusion Criteria: Patient that have suffered a MI, both Non-ST elevation MI and ST elevation MI and can be randomized within 14 days of MI with no signs of heart failure and a left ventricular ejection fraction>40%.

Main Exclusion Criteria: Any indication or contraindication for BB treatment other than secondary prevention according to the treating cardiologist

Primary study endpoint:

• The composite of all-cause mortality, recurrent MI, revascularisation with PCI or CABG, ischemic stroke, incident heart failure, or malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin.

Key secondary endpoints to be included in the main publication:

* Each of the components of the primary endpoint, i.e.: All-cause mortality, recurrent MI, revascularisation with PCI or CABG, ischemic stroke, incident heart failure, malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin.
* To study whether oral beta-blocker therapy increases the risk of hospitalization for 2 or 3rd degree AV-block, or implantation of pacemaker
* To assess clinical outcomes linked to beta-blocker therapy in the following subgroups:

age (> vs <70 years), sex (men vs. women), beta-blocker dosage, STEMI vs. NSTEMI, LVEF subgroups (preserved vs. mid-range), country, hypertension and diabetes.

Other secondary endpoints are described in the Statistical Analysis Plan and under "Outcome Measures".

Other secondary objectives (for BETAMI-DANBLOCK substudies unless specified otherwise):

* To study whether oral beta-blocker therapy reduces the risk of cardiovascular death compared to no such therapy
* To study whether oral beta-blocker therapy reduces the risk of stable and unstable angina compared to no such therapy
* To study whether oral beta-blocker therapy reduces the risk of atrial fibrillation, atrial flutter or other tachyarrhythmias compared to no such therapy
* To study whether oral beta-blocker therapy increases the risk of hospitalization for chronic obstructive pulmonary disease, asthma or peripheral artery disease.
* To study whether oral beta-blocker therapy increases the risk of hospitalization or outpatient visit for new-onset or dysregulated diabetes (DANBLOCK only)
* To study whether oral beta-blocker therapy affects the following patient related outcomes: Quality of life, angina, dyspnoea, anxiety, depression, sexual dysfunction or sleep disorders.
* To conduct cost-utility analysis in relation to quality of life and a health economic evaluation including drug use, health care utilization, employment, income, and benefit take-up
* To describe beta-blocker dosage and adherence
* To assess study safety

Safety endpoints:

The following safety endpoints will be reported in the main publication:

* Primary safety endpoint: A composite of all-cause mortality, recurrent MI, incident HF, malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin at 30 days following randomization
* Other safety endpoint: All-Cause Mortality: A table of all deaths within the follow-up period
* Other safety endpoint: Suspected Unexpected Serious Adverse Reaction (SUSARs): A table of all SUSARs within the follow-up period with number and frequency in each group. Reported by local investigators and obtained from the study databases.

All serious adverse events, including potential endpoints, are captured in the study database to be used for safety assessments and are reported continuously to regulatory authorities.

Sample Size: A total of approximately 2760 patients will be recruited and randomized 1:1 to BB treatment (type and dosage according to treating physician) or no BB treatment. Treatment must be initiated within 14 days of MI.

Sample size considerations: The study is event driven and a power calculation for the combined DANBLOCK-BETAMI trial has been performed in which 950 events will provide a power of 80% to detect a true treatment effect equal to a hazard ratio of 1.2 for no beta-blocker therapy.

Location: All departments of cardiology in Denmark are invited to participate. All patients admitted to hospital for MI will be screened for in- and exclusion criteria and contacted if eligible.

Treatment Duration: Estimated (non) treatment duration of a minimum of 6 months and a maximum of 6.25 years (anticipated).

Follow-up: Patients will be followed from the randomization date until end of follow-up.

Intervention and dosage of BB treatment: The intervention will be active treatment with BB, type and dosage according to treating cardiologist choice and control will be standard care (without BB treatment). The treating cardiologist is recommended to use the highest dose deemed tolerable for the patient at the time of randomization. Dosage, adherence and cross-over will be monitored through linkage to the Danish Register of Medical Product Statistics.

Original sample size considerations: Assuming a hazard ratio of 1.2 for the non-treated group compared to the treated the DANBLOCK trial has 80% power to detect this effect with an accumulation of 900 events of the primary endpoint. With approximately 3570 patients randomized the investigators expect to reach 900 events within the study period.

Statistical Analysis: Please see the Statistical Analysis Plan.

Data Safety Monitoring Board (DSMB): This committee consisting of two senior cardiologists and one trial-science statistician will overview safety and will have access to unblinded data. They will formally review the accumulating data every 6 months throughout the study period to ensure there is no avoidable increased harm to patients. The DSMB may recommend trial termination due to excess risk associated with no treatment with BB.

Recruitment: All patients admitted to hospital for MI will be screened for in- and exclusion criteria and contacted if eligible. Logistics of identifying and contacting the patients will be organized locally; some hospitals will randomize patients before discharge, others will contact patients after discharge. Patients will be randomized 1:1.

Publication policy: On study completion the results will be submitted for publication in an international medical journal. The results of this study will also be submitted to the Competent Authority and the Ethics Committee according to EU and Danish regulations.

Furthermore, a joint analysis of the data from BETAMI-DANBLOCK with the REDUCE (NCT03278509), CAPITAL-RCT (NCT01155635), and REBOOT (NCT03596385) trials will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction > 40%
* Myocardial infarction (MI) within previous two weeks

The diagnosis of acute MI must meet the Universal European Society of Cardiology (ESC) definition of MI

Exclusion Criteria:

* Clinical evidence of heart failure at the time of discharge
* Pregnancy or of child bearing age not using safe anticonception throughout the study period
* Lack of signed informed consent and expected cooperation during follow-up
* Any medical condition where beta blocker treatment is indicated according to the treating physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2760 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2035-12-10 (Estimated)

PRIMARY OUTCOMES:
A composite of all-cause mortality, recurrent MI, revascularisation with PCI or CABG, ischemic stroke, incident heart failure, or malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin. | Estimated follow-up min 6 months - max 6.25 years
  Time to the composite of all-cause mortality, recurrent MI, revascularisation with PCI or CABG, ischemic stroke, incident heart failure, or malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiag origin on an intention to treat analysis. The composite outcome will be assessed through nationwide registries and adjudicated by an independent Clinical Endpoint Adjudication Committee.

SECONDARY OUTCOMES:
Recurrent myocardial infarction | Estimated follow-up min 6 months - max 6.25 years
  Key secondary endpoint. Assessed through nationwide registries.
All-cause mortality | Estimated follow-up min 6 months - max 6.25 years
  Key secondary endpoint. Assessed through nationwide registries.
Malignant ventricular arrhythmias | Estimated follow-up min 6 months - max 6.25 years
  Key secondary endpoint. Assessed through nationwide registries.
Incident heart failure (diagnosed at hospitalization or at out-patient visits) | Estimated follow-up min 6 months - max 6.25 years
  Key secondary endpoint. Assessed through nationwide registries.
Unplanned coronary revascularization | Estimated follow-up min 6 months - max 6.25 years
  Key secondary endpoint. Assessed through nationwide registries.
Ischemic stroke | Estimated follow-up min 6 months - max 6.25 years
  Key secondary endpoint. Assessed through nationwide registries.
Resuscitated cardiac arrest of cardiac origin | Estimated follow-up min 6 months - max 6.25 years
  Key secondary endpoint. Assessed through nationwide registries.
Cardiovascular mortality | Estimated follow-up min 6 months - max 6.25 years
  Assessed through nationwide registries.
Hospitalization for stable and unstable angina pectoris | Estimated follow-up min 6 months - max 6.25 years
  Assessed through nationwide registries.
Hospitalization for atrial fibrillation, atrial flutter or other tachyarrhythmias | Estimated follow-up min 6 months - max 6.25 years
  Assessed through nationwide registries.
Hospitalization for bradycardia, AV-block, syncope, or need for pacemaker | Estimated follow-up min 6 months - max 6.25 years
  Assessed through nationwide registries.
Hospitalization for asthma and chronic obstructive pulmonary disease symptoms | Estimated maximal follow-up 6 months - 6.25 years
  Assessed through nationwide registries.
Hospitalization or outpatient visit for peripheral artery disease | Estimated follow-up min 6 months - max 6.25 years
  Assessed through nationwide registries.
Hospitalization or outpatient visit for new-onset or dysregulated diabetes (DANBLOCK only) | Estimated follow-up min 6 months - max 6.25 years
  Assessed through nationwide registries.
Angina symptoms | E-questionnaires will be administered at inclusion, 3, 12 and 24 months
  Canadian Cardiovascular Society (CCS) grading of angina pectoris.
Exercise capacity (DANBLOCK only) | At the beginning of cardiac rehabilitation (within approximately 4 weeks after randomization) and at the end of cardiac rehabilitation (approximately 6-12 weeks after beginning of rehabilitation)
  Data on exercise capacity (VO2peak) will measured before and after rehabilitation and recorded in the Danish Cardiac Rehabilitation database.
Blood pressure control (DANBLOCK only) | At the beginning of cardiac rehabilitation (within approximately 4 weeks after randomization) and at the end of cardiac rehabilitation (approximately 6-12 weeks after beginning of rehabilitation)
  Data on blood pressure (systolic and diastolic) will measured before and after cardiac rehabilitation and recorded in the Danish Cardiac Rehabilitation database
Quality of life measure | E-questionnaires will be administered at inclusion, 3, 12 and 24 months
  EQ5D (a measure of health-related quality of life that can be used in a wide range of health conditions and treatments)
Measures of depression and anxiety | E-questionnaires will be administered at inclusion, 3, 12 and 24 months
  HADS (Hospital Anxiety and Depression Scale)
Measures of sexual dysfunction | E-questionnaires will be administered at inclusion, 3, 12 and 24 months
  The International Index of Erectile Function (IIEF) and Female Sexual Function Index (FSFI)
Measures of sleeping disorder | E-questionnaires will be administered at inclusion, 3, 12 and 24 months
  Bergen insomnia Scale
Adherence to the prescribed dosage of beta-blocker | Estimated follow-up min 6 months - max 6.25 years
  Assessed through nationwide registries.
Cost-utility analysis in relation to quality of life and a health economic evaluation including drug use, health care utilization, employment, income, and benefit take-up | Estimated follow-up min 6 months - max 6.25 years
  Assessed through nationwide registries and study database

CONTACTS AND LOCATIONS:
Overall Officials: Eva IB Prescott, MD, DMsC, Principal Investigator — Bispebjerg Frederiksberg University Hospital; Anna Meta D Kristensen, MD, Study Chair — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Bispebjerg Hospital, Dept. of Cardiology Y builing 67, 1.floor, Bispebjerg Bakke 23, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Munkhaugen J, Kristensen AMD, Halvorsen S, Holmager T, Olsen MH, Bakken A, Sehested TSG, Ruddox V, Maeng M, Vikenes K, Jensen SE, Steigen T, Lambrechtsen J, Jortveit J, Bovin A, Schirmer H, Christiansen MK, Wiseth R, Mikkelsen D, Larsen AI, Lyngby Kjaergaard C, Andresen K, Gustafsson I, Tuseth V, Larsen ML, Deeg PS, Veien K, Bohmer E, Botker HE, Brattrud AO, Bronnum-Schou J, Pettersen AR, Bang LE, Oie E, Engstrom T, Borg EB, Kristensen K, Nymo SH, Gislason G, Vethe NT, Abdulla JAM, Dammen T, Mouridsen MR, Bendz B, Bertelsen MLN, Hove JD, Schierbeck L, Snoer M, Davidsen C, Egholm G, Thomsen KK, Jadou G, Poenaru M, Krarup NT, Bottcher M, Staehr PB, Zwisler AD, Edvardsen T, Torp-Pedersen C, Otterstad JE, Lange T, Fagerland MW, Atar D, Prescott E; BETAMI-DANBLOCK Investigators. Beta-Blockers after Myocardial Infarction in Patients without Heart Failure. N Engl J Med. 2025 Nov 13;393(19):1901-1911. doi: 10.1056/NEJMoa2505985. Epub 2025 Aug 30. PMID 40888716
- [Derived] Kristensen AMD, Bovin A, Zwisler AD, Cerquira C, Torp-Pedersen C, Botker HE, Gustafsson I, Veien KT, Thomsen KK, Olsen MH, Larsen ML, Nielsen OW, Hildebrandt P, Foghmar S, Jensen SE, Lange T, Sehested T, Jernberg T, Atar D, Ibanez B, Prescott E. Design and rationale of the Danish trial of beta-blocker treatment after myocardial infarction without reduced ejection fraction: study protocol for a randomized controlled trial. Trials. 2020 May 23;21(1):415. doi: 10.1186/s13063-020-4214-6. PMID 32446298

DOCUMENTS (2):
  • Study Protocol (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03778554/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03778554/SAP_002.pdf